CLINICAL TRIAL: NCT06545175
Title: Extracellular Vesicle-enriched Secretome Fraction (VSF1.01) for the Reduction of Cochlear Implant Surgery Related Trauma (ESCRT). An Open-label Monocentric Phase I/IIa Clinical Trial to Investigate the Safety of Intracochlear Application of VSF1.01 Enriched With hUC-MSC-EVs in Patients Receiving Cochlear Implantation.
Brief Title: Intracochlear Application of VSF1.01 for the Reduction of Cochlear Implant Surgery Related Trauma
Acronym: ESCRT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-512498-29-00
Record Dates: First submitted 2024-07-16; First posted 2024-08-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intracochlear treatment with VSF1.01 (Experimental)
  Interventions: Drug: Intracochlear application of VSF1.01

INTERVENTIONS:
Drug: Intracochlear application of VSF1.01 — During cochlear implant operation, patients receive intracochlear VSF1.01 prior to insertion of the electrode array.

SUMMARY:
The goal of this clinical trial is to assess the safety of intracochlear application of VSF1.01 for the reduction of cochlear implant surgery related trauma in patients with profound hearing loss with or without non-functional residual hearing in low frequencies and cochlear implantation.

The main questions it aims to answer are:

Primary objective:

Safety of intracochlear application of VSF1.01 in patients receiving cochlear implantation

Secondary objectives:

Effectiveness on

1. neural responses of auditory nerve
2. speech understanding
3. hearing thresholds
4. electrode impedances

During cochlear implant operation, patients receive as adjuvant treatment intracochlear VSF1.01 prior to insertion of the electrode array.

Cochlear implantation is conducted according to the clinical standard at the investigational site.

ELIGIBILITY:
Inclusion Criteria:

* Men, women, inter/diverse aged ≥ 18 years

  * Women without childbearing potential defined as follows:

    * at least 6 weeks after surgical sterilization by bilateral tubal ligation or bilateral oophorectomy or
    * hysterectomy or uterine agenesis or
    * ≥ 50 years and in postmenopausal state > 1 year or
  * Women of childbearing potential:

    * who are practicing sexual abstinence (periodic abstinence and withdrawal are not acceptable) or
    * who have sexual relationships with female partners only and/or with sterile male partners or
    * who are sexually active with fertile male partner, have a negative pregnancy test during screening and agree to use reliable methods of contraception from the time of screening until end of the clinical trial.
* Signed written informed consent from subjects capable of understanding all information and to give full informed consent
* Functional deaf patients (profound hearing loss with or without non-functional residual hearing in the low frequencies i.e. 125 Hz: 45 dB - 95 dB; 250 Hz: 50 dB - 105 dB; 500 Hz: 55 dB - 110 dB; 750 Hz and higher: 65 dB or below) that are candidates for cochlear implantation

Exclusion Criteria:

* Patients with prior ear surgery
* Patients with inner ear malformations
* Patients with acute or chronic otitis media
* Patients with keloid disorder
* Comorbidities concerning the central nervous system
* Malignancies of any type
* Kidney disease with elevated blood values: creatinine >1.5x above upper limit of normal (ULN), eGFR or creatinine clearance 59 mL/min/1.73 m2 (grade ≥2, CTCAE v5.0)
* Liver disease with elevated blood values: bilirubin >1.5x ULN, AST/ALT >3.0x ULN, ALP and y-GT >2.5x ULN, LDH >ULN, international normalized ratio (INR) >1.5-2.5x baseline if on anticoagulation, albumin <3 g/dL (grade ≥2, CTCAE v5.0)
* Suspected or verified pregnancy or breastfeeding
* Hypersensitivity to any of the components of the medications used (such as Ringer's Lactate (excipient); any residuals from cell culture or raw materials used for pharmaceutical upstream and downstream processing to generate VSF1.01 (i.e. alpha-Modified Eagle Medium (αMEM), Dulbecco's MEM (DMEM), pooled human platelet lysate (pHPL), human serum albumin (HSA), Dipeptiven, phosphate buffered saline (PBS), animal origin free recombinant enzyme (TrypLETM Select))
* Participation in another clinical trial (other investigational drugs or devices at the time of enrolment or within 30 days prior to enrolment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate and severity of (serious) adverse events | Continuously from start to end of study [Start: IMP treatment (day 0), end of the study (Follow-up 5)], assessed up to approximately 6 months
  Recording and documentation of number and severity of (serious) adverse events

SECONDARY OUTCOMES:
Evaluation of eCAP growth function | Continuously from start to end of study [Start: IMP treatment (day 0), end of the study (Follow-up 5)], assessed up to approximately 6 months
  Assessment of effectiveness on neural responses of auditory nerve by measuring electrically evoked compound action potential (eCAP; eCAP growth function)
Evaluation of speech perception | From Day 1 (FU 1) to end of study (FU 5), assessed up to approximately 6 months
  Assessment of effectiveness on speech understanding by measuring speech perception (in quiet and in noise) by HSM 10dB SNR/5dB SNR, FBM, OLSA 50%
Measurement of air and bone conduction | At Screening/baseline and from Day 1 (FU 1) to end of study (FU 5), assessed up to approximately 6 months
  Assessment of effectiveness on hearing thresholds by measuring air and bone conduction from 125 Hz - 16,000 Hz by pure tone audiometry
Measurement of impedance levels | From Day 0 to end of study (FU 5), assessed up to approximately 6 months
  Assessment of effectiveness on electrode impedances by determination of impedance levels (as measure to rule out pathological levels and as part of clinical routine)

CONTACTS AND LOCATIONS:
Overall Officials: Nils K. Prenzler, PD DR., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Dept. of Otorhinolaryngology, Hanover, Germany